CLINICAL TRIAL: NCT01482806
Title: Online Treatments for Mood and Anxiety Disorders in Primary Care
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bruce Rollman, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH093501 (NIH)
Record Dates: First submitted 2011-11-22; First posted 2011-12-01 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Depression; Generalized Anxiety Disorder; Panic Disorder
Keywords: Depression; Anxiety; Primary care; Cognitive Behavioral Therapy; Internet; Support groups; Technology assisted
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computerized CBT + Internet Support Group (Experimental): Guided patient access to Beating the Blues plus access to a moderated ISG where patients will be able to communicate confidentially to receive and provide advice and peer-support from other study participants (CCBT+ISG; N=300).
  Interventions: Behavioral: CCBT+ISG/Collaborative Care
- Computerized CBT Alone (Experimental): Guided patient access to Beating the Blues, a proven-effective, on-line 8-session CCBT program approved for use in the United Kingdom (CCBT-alone; N=300).
  Interventions: Behavioral: CCBT/Collaborative Care
- Usual Care (No Intervention): Primary care physicians' "usual care" for mood and anxiety disorders (UC; N=100).

INTERVENTIONS:
Behavioral: CCBT+ISG/Collaborative Care — Guided patient access to the Beating the Blues CCBT program plus access to a moderated ISG where patients will be able to communicate confidentially to receive and provide advice and peer-support from other study participants
  These interventions will be delivered as part of a collaborative care intervention provided in concert with their usual source of primary care.
  Patients will also have the option of pharmacotherapy for their mood and/or anxiety disorder and referral to a community mental health specialist per their preference.
  Arms: Computerized CBT + Internet Support Group
Behavioral: CCBT/Collaborative Care — Guided patient access to the Beating the Blues CCBT program.
  This interventions will be provided as part of a collaborative care intervention provided in concert with their usual source of primary care.
  Patients will also have the option of pharmacotherapy for their mood and/or anxiety disorder and referral to a community mental health specialist per their preference.
  Arms: Computerized CBT Alone

SUMMARY:
Depression and anxiety are common in primary care practice and are associated with substantial reductions in health-related quality of life. This Project will test the comparative effectiveness of two on-line treatments for these conditions provided through the context of a Collaborative Care program: (1) moderated access to a proven-effective computerized cognitive behavioral therapy (CCBT) program; versus (2) moderated access to CCBT plus an Internet support group (CCBT+ISG). The Project will also compare the effectiveness of these treatments to PCPs' "usual care" for these conditions, and evaluate the adoption and maintenance of CCBT+ISG by practices following the conclusion of the trial to provide a greater understanding of how to best scale the delivery of these interventions into a variety of primary care settings.

DETAILED DESCRIPTION:
Depression and anxiety are prevalent in primary care practice, associated with substantial reductions in health-related quality of life (HRQoL), and generate a significant excess of morbidity. In response, dozens of trials have demonstrated the greater effectiveness of "Collaborative Care" for these conditions vs. primary care physicians' usual care. Yet for a variety of reasons, these models have not been widely implemented. Therefore, an urgent need remains to develop and test more scalable, powerful, and innovative versions of Collaborative Care while simultaneously developing a greater understanding of how best to provide these interventions through primary care where the majority of depressed and anxious patients seek treatment.

Thousands of web sites provide medical information and the number of Internet support groups (ISG) where the public can exchange information about treatments is proliferating. Still, clinical trials have not established the benefits of utilizing the Internet in this manner. Concurrent with these developments, several computerized cognitive behavioral therapy (CCBT) programs have been proven effective at treating patients with mood and anxiety disorders and used by hundreds of thousands of patients outside the U.S. Yet CCBT remains little utilized inside the U.S., and no trials have incorporated CCBT into a Collaborative Care intervention or examined the effectiveness of combining CCBT with an ISG for these disorders.

We propose a 4-year comparative effectiveness trial that will randomize 700 primary care patients aged 18-75 who have at least a moderate level of mood and/or anxiety symptoms and reliable access to both the Internet and e-mail to either: (1) guided patient access to Beating the Blues, a proven-effective on-line CCBT program (CCBT-alone; N=300); (2) guided patient access to Beating the Blues plus access to a moderated ISG (CCBT+ISG; N=300); or (3) their PCP's "usual care" (N=100). Our primary hypothesis is that patients in our CCBT+ISG arm will report a clinically meaningful 0.30 effect size (ES) or greater improvement in HRQoL on the SF-12 MCS compared to patients in our CCBT-alone arm at 6-months follow-up, and we will monitor patients for an additional 6 months to evaluate the durability of our interventions. Our secondary hypothesis is that CCBT-alone patients will report a 0.50 ES or greater improvement in HRQoL on the SF-12 MCS versus "usual care" at 6-months follow-up. To better understand how online mental health treatments are best provided through primary care, we will also evaluate: (a) their effectiveness across and within age strata; (b) their cost-effectiveness; (c) how patients utilize the components of our interventions; (d) patient subgroups for whom our interventions may be particularly effective; and (e) the adoption and maintenance of our interventions by practices following the Intervention Phase of the Project. Study findings are likely to have profound implications for transforming the way mental health conditions are treated in primary care and focus further attention to the emerging field of e-mental health by other U.S. investigators.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 Years of age.
* Current major depression, panic, and/or generalized anxiety disorder on PRIME-MD.
* At least a moderate level of mood and/or anxiety symptoms (PHQ-9 ≥ 10 or a GAD-7 ≥ 10).
* Not receiving treatment for a mood or anxiety disorder from a mental health specialist.
* Has a telephone, e-mail address, and reliable access to the Internet.
* Stable medical condition and life expectancy greater than one year.

Exclusion Criteria:

* Active suicidal ideation or psychotic disorder.
* History of bipolar disorder.
* Alcohol dependence or other substance abuse disorder within the past three months.
* Plans to leave present source of care over the following year.
* Non-English speaking, illiterate, or having a visual or auditory barrier limiting ability to participate in telephone assessments, interventions, or provide signed, informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
SF-12 MCS | 6-Month Follow-up
  The investigators will assess all study patients' mental health-related quality of life (HRQoL) on the SF-12 MCS via telephone at 6-months follow-up, and we will monitor patients for an additional 6 months to evaluate the durability of our interventions.

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression | 6-Months
  The investigators will assess all study patients' mood symptoms using the HRS-D via telephone at 6-months follow-up, and we will monitor patients for an additional 6 months to evaluate the durability of our interventions.
Hamilton Rating Scale for Anxiety | 6-Months
WHO Health and Work Performance Questionnaire | 6-Months
Health Services Utilization and Costs | 12-Months
Attitudes to Computerized CBT | 6-Months
Computerized CBT and Internet Support Group Usage | 12-Months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Rollman, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Rollman BL, Herbeck Belnap B, Rotondi AJ. Internet support groups for health: ready for the Affordable Care Act. J Gen Intern Med. 2014 Nov;29(11):1436-8. doi: 10.1007/s11606-014-2884-z. No abstract available. PMID 24817281
- [Background] Herbeck Belnap B, Schulberg HC, He F, Mazumdar S, Reynolds CF 3rd, Rollman BL. Electronic protocol for suicide risk management in research participants. J Psychosom Res. 2015 Apr;78(4):340-5. doi: 10.1016/j.jpsychores.2014.12.012. Epub 2014 Dec 27. PMID 25592159
- [Background] Jonassaint CR, Gibbs P, Belnap BH, Karp JF, Abebe KK, Rollman BL. Engagement and outcomes for a computerised cognitive-behavioural therapy intervention for anxiety and depression in African Americans. BJPsych Open. 2017 Jan 2;3(1):1-5. doi: 10.1192/bjpo.bp.116.003657. eCollection 2017 Jan. PMID 28058109
- [Background] Cavanagh K, Herbeck Belnap B, Rothenberger SD, Abebe KZ, Rollman BL. My care manager, my computer therapy and me: The relationship triangle in computerized cognitive behavioural therapy. Internet Interv. 2017 Nov 6;11:11-19. doi: 10.1016/j.invent.2017.10.005. eCollection 2018 Mar. PMID 30135755
- [Background] Rollman BL, Herbeck Belnap B, Abebe KZ, Spring MB, Rotondi AJ, Rothenberger SD, Karp JF. Effectiveness of Online Collaborative Care for Treating Mood and Anxiety Disorders in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Jan 1;75(1):56-64. doi: 10.1001/jamapsychiatry.2017.3379. PMID 29117275
- [Background] Geramita EM, Herbeck Belnap B, Abebe KZ, Rothenberger SD, Rotondi AJ, Rollman BL. The Association Between Increased Levels of Patient Engagement With an Internet Support Group and Improved Mental Health Outcomes at 6-Month Follow-Up: Post-Hoc Analyses From a Randomized Controlled Trial. J Med Internet Res. 2018 Jul 17;20(7):e10402. doi: 10.2196/10402. PMID 30021711
- [Background] Jonassaint CR, Belnap BH, Huang Y, Karp JF, Abebe KZ, Rollman BL. Racial Differences in the Effectiveness of Internet-Delivered Mental Health Care. J Gen Intern Med. 2020 Feb;35(2):490-497. doi: 10.1007/s11606-019-05542-1. Epub 2019 Nov 19. PMID 31745855
- [Background] Rollman BL, Brent DA. Phonotype: a New Taxonomy for mHealth Research. J Gen Intern Med. 2020 Jun;35(6):1881-1883. doi: 10.1007/s11606-019-05407-7. Epub 2019 Nov 8. No abstract available. PMID 31705476
- [Derived] Rotondi AJ, Belnap BH, Rothenberger S, Feldman R, Hanusa B, Rollman BL. Predictors of Use and Drop Out From a Web-Based Cognitive Behavioral Therapy Program and Health Community for Depression and Anxiety in Primary Care Patients: Secondary Analysis of a Randomized Controlled Trial. JMIR Ment Health. 2024 Jan 17;11:e52197. doi: 10.2196/52197. PMID 38231552
- [Derived] Morone NE, Herbeck BB, Huang Y, Abebe KZ, Rollman BL, Jonassaint CR. The Impact of Optimism and Pain Interference on Response to Online Behavioral Treatment for Mood and Anxiety Symptoms. Psychosom Med. 2021 Nov-Dec 01;83(9):1067-1074. doi: 10.1097/PSY.0000000000000980. PMID 34267085
- See also: Related Info — http://insideupmc.blogspot.com/2012/12/trial-explores-using-internet-to-treat.html